CLINICAL TRIAL: NCT03928964
Title: Pronostic Assessment of Mortality Among Locally Advanced or Metastatic Renal Cell Carcinoma Patients After First Line Treatment : Multicenter Prospective Cohort Study With Historic Medical Data
Brief Title: MEtatastic Renal Carcinoma LINes
Acronym: MERLIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2017/342
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis of this study are as follows:

* Prognostic evaluation of patients based on an integrative model provides better assessment of overall survival, and thus improves setting of care goals.
* In a routine care population, antitumour drugs may have a significant impact on overall survival through their targeted antitumor effect, but also through their toxicity profile and their impact on comorbidities.
* The optimization of patient support (supportive care, drug tolerance monitoring) can have an impact on the prognosis.

ELIGIBILITY:
Inclusion criteria:

1. Patients with locally advanced or metastatic renal cell carcinoma
2. Whose first-line treatment included at least one anti-angiogenic agent (tyrosine kinase inhibitor or monoclonal antibodies) and / or an mTOR inhibitor;
3. Whatever was the overall ECOG-PS score (Eastern Cooperative Oncology Group Performance Status) at treatment initiation time
4. With first-line treatment carried out between 2007 and June 2016.

Exclusion criteria:

1. Patient previously treated with only one cytokine (Interferon α2a, high-dose interleukin-2)
2. Refusal of processing of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic renal cell carcinoma, whose first-line treatment included at least one anti-angiogenic agent (tyrosine kinase inhibitor or monoclonal antibodies) and / or an mTOR inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival after the first line of treatment | year 11
  Time elapsed between initiation date for 2nd line treatment et the date of death, whatever the cause.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Rousseau, MD, Principal Investigator — Henri Mondor University Hospital
Locations (8):
- France (8):
  - CHU de Besançon, Besançon
  - Hôpital Henri Mondor, Créteil
  - Hôpital Nord Franche-Comté Montbéliard, Montbéliard
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint-Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital d'Instruction des Armées de Bégin, Saint-Mandé

IPD SHARING:
Plan to Share IPD: No